CLINICAL TRIAL: NCT00325845
Title: Efficacy and Safety of Intra-Articular Synvisc Injections as Treatment of Painful Lumbar Facet Joint Arthrosis
Brief Title: Synvisc Injections for Lumbar Facet Joint Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheltering Arms Physical Rehabilitation Hospitals (Other)
Collaborators: Genzyme, a Sanofi Company (Industry); Virginia Commonwealth University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G050253
Record Dates: First submitted 2006-05-12; First posted 2006-05-15 (Estimated); Last update posted 2006-09-13 (Estimated); Status verified 2006-09

CONDITIONS: Joint Pain
Keywords: Investigational; Therapeutic; Efficacy; Safety; Outcomes; Lumbar facet joint arthrosis; Lumbar facet joint arthropathy
MeSH Terms: conditions — Arthralgia

INTERVENTIONS:
Procedure: Synvisc viscosupplementation

SUMMARY:
The objective of this investigation is to evaluate the safety and efficacy of viscosupplementation in treating symptomatic lumbar facet joint arthropathy. The intended use of the device (Synvisc) is to alleviate pain and improve function in patients with painful lumbar facet joint arthrosis by intra-articular injection into the involved joint.

DETAILED DESCRIPTION:
Patients will enter the study once the putatively painful joint or joints have been confirmed by single blind, double local-comparative anesthetic blockade. The joint(s) suspected by historical features and physical examination will be injected under fluoroscopic guidance with contrast-enhancement confirming intra-articular placement. The initial injectate will be 1cc of 2% xylocaine. Single diagnostic lumbar facet joint injections carry a false positive rate of 38%. In order to maximize the specificity of the diagnostic injections a second 1cc injection of a longer-acting local anesthetic, 0.5% marcaine, will be performed on all patients reporting clinically significant pain reduction (> 75% VAS reduction from pre-injection baseline) within 10-15 minutes after the xylocaine injection. This second diagnostic injection will be completed upon return of the patient's pain back to baseline (no sooner than 3 days after the initial diagnostic injection). A true positive response will be defined as > 50% VAS reduction after the second injection. Patients will then undergo 2 IA Synvisc injections into the painful facet joint(s). An initial IA injection of 1.0cc (or a volume, not to exceed 1.0cc, accepted by the joint upon reaching a capsular endpoint) of Synvisc (1cc, 10mg/ml) will be injected into the painful joint(s) 7 days after the second diagnostic injection after the baseline pain has returned. A 2nd injection will then be performed 10 days after the initial injection. A 3rd injection may be offered to patients not satisfied with the results obtained with the first 2 Synvisc injections. A 2.0cc vial of Synvisc per patient will be shipped including other trial materials to the investigator for implementation. A fluid dispenser connector will allow direct dispensation of 1.0cc of Synvisc from the pre-packaged 2.0cc unmarked vial. Outcome measurement tools will include Visual Analogue Scale, Oswestry Disability Questionnaire, SF-36, lumbar spine range of motion (ROM), sitting and walking tolerance, analgesic usage, and patient satisfaction. Data will be collected at baseline, at 7-10 days after the second Synvisc injection, and at 1, 3, 6, and 12 month follow up (after the final Synvisc injection) visits. For example, patient X will undergo an initial 2 Synvisc injections and then be evaluated in the office 7 days later. If the patient experiences significant benefit, no other injections will be pursued. However, if a therapeutic benefit is achieved but is not satisfactory to the patient, a 3rd Synvisc injection will be performed within 3 days. A side effect and complications questionnaire will be completed by each patient within 30 minutes, 24 hours, and 72 hours after each injection (including diagnostic injections).

ELIGIBILITY:
Inclusion Criteria:

1. Ongoing axial lumbar pain, greater than any lower limb pain if present, for > 3 months duration.
2. No improvement despite 6-8 weeks of physical therapy (PT), oral nonsteroidal anti-inflammatory drugs (NSAIDs), relative rest, and activity modification.
3. Radiographic evidence of facet joint arthrosis on advanced imaging studies defined as joint capsule hypertrophy, osteophyte formation, joint space narrowing, irregularity of joint contours, subchondral sclerosis, and synovial cyst formation.
4. Age 30 years or older.
5. Positive double, local comparative anesthetic diagnostic block injections at one unilateral or bilateral joint(s).

Exclusion Criteria:

1. Pregnancy.
2. Active or remote history of spinal malignancy.
3. Active infection.
4. Blood dyscrasias/coagulopathy.
5. Unwillingness to follow through with follow up evaluations.
6. Negative response to all diagnostic facet joint injections.
7. Application for/currently receiving worker's compensation.
8. Allergy to avian products.
9. Allergy to prior viscosupplementation products.
10. Prior viscosupplementation of lumbar facet joints.
11. Improper intra-articular needle placement at time of Synvisc injection.
12. Painful bilateral or multi-level facet joint arthropathy.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2006-05; Study Completion 2008-05

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) for baseline pain (best, worst, average) and pain while walking
Oswestry Disability Questionnaire
Short Form 36-Item (SF-36)
Standing/walking tolerance (defined as time patient can sit for before pain level reaches baseline or distance walked before pain reaches baseline)

SECONDARY OUTCOMES:
Analgesic usage
Lumbar range of motion
Patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Michael J DePalma, MD, Principal Investigator — Sheltering Arms Physical Rehabilitation Hospitals; Virginia Commonwealth University
Locations (1):
- Sheltering Arms Spine and Sport Center; St. Mary's Hospital, Richmond, Virginia, United States